## **Informed consent**

México CDMX. March 3<sup>th</sup> 2016

Effect of Acute or Chronic Ingestion of Sucralose on Serum Insulin in Young and Healthy Adults: A Randomized, Double-Blind, Placebo-Controlled Trial.

This document was sent in order to inform Dr. Guillermo Melendez Mier the protocol approval by the Investigation Ethics Committee of the General Hospital of Mexico. This document establish the confidence of the study methodology, according to the Helsinski declaration, ensuring the health, welfare and rights of participants.





Document number CE/091/16

Mexico City, march 3th, 2016

**DR. GUILLERMO MELENDEZ MIER** Investigation departament chief.

Dear Dr. Melendez

The Investigation Ethics Committee wants to make of your knowledge the approval of the protocol named: "SERUM INSULIN AN GLUCOSE RESPONSE AFTER ACUTE AND CHRONIC SUCRALOSE INGESTION IN HEALTHY PATIENTS WITH VARIABLE BODY MASS INDEX".

The last version of the protocol has been approved by the Investigation ethics committee this march the  $\mathbf{1}^{\text{st}}$  of the present year, in order to be acomplished by your coordination at the investigation departament.

At the same time, the informed consent has been approved to be used in this cinical trial.

Every time the protocol is changed, the modifications should be submitted to this committee for an approval.

The committee will be greatful for recieving the renewal of this protocol authorization with a development summary of the reserch that you are in charge of annexed.

Once the study is completed, we kindly request for a results obtained report.

Yours cordially,

DRA! ESTHELA GARCIA ELVIRA

Investigation Ethics Committee president.

"At the forefront in the care of life"

